CLINICAL TRIAL: NCT02478372
Title: Patient Controlled Epidural Analgesia Versus Local Infiltration Analgesia Following Knee Arthroplasty Within an Enhanced Recovery Programme - a Randomised Controlled Trial
Brief Title: Patient Controlled Epidural Analgesia Versus Local Infiltration Analgesia Following Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Jubilee National Hospital (Other Government)
Collaborators: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/ORTH/01
Record Dates: First submitted 2015-04-02; First posted 2015-06-23 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis
Keywords: local infiltration analgesia; Epidural; Enhanced Recovery; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis | interventions — Levobupivacaine; Bupivacaine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Controlled Epidural (PCEA) (Active Comparator): A lumbar epidural was sited using a side-directed technique towards the side of surgery following establishment of the spinal blockade. Following the completion of the operation, patients received 4ml of 0.25% levobupivacaine prior to leaving the operating room. Thereafter they were connected to a PCEA pump (McKinley 545) with no background infusion. Patients could self-medicate with a bolus 2ml of 0.125% bupivacaine via the PCEA system with a lockout time of 15 minutes to control their pain until the following morning (post-operative day one) when it was stopped. Nurse-administered rescue top-ups of 4ml of 0.25% levobupivacaine were available for insufficient analgesia. The epidural catheter was removed on the morning of post-operative day two (POD2).
  Interventions: Drug: Patient Controlled Epidural (PCEA)
- Local Infiltration Analgesia (LIA) (Experimental): Subcutaneous infiltration during surgery using 200ml of 0.2% plain ropivacaine. 50ml injected following bone preparation prior to implant cementation perpendicular to the posterior femur through the posterior joint capsule in 10ml aliquots. 30ml proximal to the suprapatellar pouch down to the femur.100ml spread into subcutaneous tissues including; collateral and cruciate ligaments, fatty and connective tissue on the anterior aspect of the incision. A 16 gauge epidural catheter inserted via a medial portal, 20ml was injected via the catheter following closure of wound. Post-operatively, patients received boluses of 40ml ropivacaine 0.2% via the catheter using a mechanical McKinley 595 pump 4 hours after leaving theatre, at 22:00 and 08:00 on post-operative day one.
  Interventions: Drug: Local Infiltration Analgesia (LIA)

INTERVENTIONS:
Drug: Patient Controlled Epidural (PCEA) — Following the operation, 4ml of 0.25% levobupivacaine was administered and the catheter was connected to a PCEA. Self-medication with a bolus 2ml of 0.125% bupivacaine via the PCEA system with a lockout time of 15 minutes until the following morning (post-operative day one) when it was stopped.
  Other Names: Levobupivacaine and Bupivacaine
  Arms: Patient Controlled Epidural (PCEA)
Drug: Local Infiltration Analgesia (LIA) — Subcutaneous infiltration during surgery using 200ml of 0.2% plain ropivacaine.
  Other Names: Ropivacaine
  Arms: Local Infiltration Analgesia (LIA)

SUMMARY:
The purpose of this study was to determine if the method of peri-operative analgesia used following total Knee Replacement surgery affected the progress towards rehabilitation goals and to determine whether the analgesia had any impact on long term outcomes.

DETAILED DESCRIPTION:
Enhanced Recovery Programmes (ERP) as defined by Henrik Kehlet have been established within orthopaedics within the United Kingdom in a number of centres (Malviya et al., 2011, McDonald et al., 2012, Scott et al., 2013) demonstrating improvements in patient outcomes. However as the ERP involved in all of these papers are a redesign of a number of key elements of the clinical pathway it remains unclear as to the level of significance each component may have on the patient's reported outcomes.

The use of Local Infiltration Analgesia (LIA) as the primary post-operative analgesic technique has grown in popularity in Scotland over the past 5 years (Scott et al., 2013). A number of large cohort series have concurrently reported significant improvements in early ambulation and shortened lengths of stay (Malviya et al., 2011, McDonald et al., 2012) yet it remains unclear as to whether this is due to the introduction and use of the LIA technique or the overall development of the ERP programmes.

The aim of this parallel group randomised controlled trial was to test two different methods of regional analgesia (LIA and Epidural) and their impact on attainment of predetermined rehabilitation criteria for direct discharge home and to consider the impact of each technique on long term functional status up to one year post surgery.

Epidural analgesia when utilised as post-operative analgesia is predominantly used in the format of a continuous infusion of a set volume of analgesia (+/- adjuncts such as fentanyl) resulting in both a motor and sensory blockade, which as would be expected increases with the volume infused. Ambulatory patient epidurals have been used for a number of years within maternity services which provide adequate pain relief whilst enabling the patient to be mobile (Stewart & Fernando, 2011). Therefore to provide a fairer comparison with the LIA technique the standard epidural analgesia technique within the Golden Jubilee National Hospital was adapted to a Patient Controlled Epidural Analgesia (PCEA) system with no background infusion.

The planned long term follow up period ( One year) was developed to enable greater evidence of the impact of each method on functional capacity, Patient Reported Outcome Scores (PROMS) and to monitor the incidence of adverse incidents over a longer period of time than previously published literature.

ELIGIBILITY:
Inclusion Criteria:

* All patients (age> 18years old) undergoing primary unilateral total knee arthroplasty (TKA) with a clinical diagnosis of osteoarthritis

Exclusion Criteria:

* Patients planned for uni-compartmental/bilateral or revision knee surgery patients
* Patients with a diagnosis of rheumatoid arthritis (RA)
* Patients with coagulation or anatomical defects e.g. preventing the use of spinal anaesthesia
* Known allergies to any medications within the trial
* Patients who were unable to give written informed consent
* Patients requiring pre-operative catheterisation for urinary outflow dysfunction
* Known neurological incident that would limit or make impossible early ambulation following surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A McDonald, BSc, Principal Investigator — Golden Jubilee National Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Controlled Epidural (PCEA): A lumbar epidural was sited following establishment of the spinal blockade. Following the completion of the operation, patients received 4ml of 0.25% levobupivacaine prior to leaving the operating room. Thereafter they were connected to a PCEA pump (McKinley 545) with no background infusion. Patients could self-medicate with a bolus 2ml of 0.125% bupivacaine via the PCEA system with a lockout time of 15 minutes until the following morning (post-operative day one). Nurse-administered rescue top-ups of 4ml of 0.25% levobupivacaine were available for insufficient analgesia. The epidural catheter was removed on the morning of post-operative day two (POD2).
Period: Overall Study
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Started | 121 | 121
Recieved Allocation Intervention | 109 | 113
Reviewed at Six Weeks | 108 (Routine follow up at six weeks - one patient refused to attend) | 113 (Routine follow up at six weeks)
Reviewed at One Year | 108 (Routine follow up at one year) | 107 (Routine folow up at one year - four patients did not attend, two patients died)
Completed | 108 | 107
Not Completed | 13 | 14
Not completed — Protocol Violation | 12 | 8
Not completed — Lost to Follow-up | 1 | 4
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Population: Total number of patients recruited to each arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA) | Total
Number analyzed (Participants) | 121 | 121 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10) | 68 (11) | 67 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 71 | 137
  Male | 55 | 50 | 105
Region of Enrollment [Number; unit: participants]
  United Kingdom | 121 | 121 | 242
Body Mass Index [Mean (Standard Deviation); unit: kilogrammes per meter squared] — Weight (kilogrammes) divided by height squared (meters)
  kilogrammes per meter squared | 31 (8) | 31 (8) | 31 (8)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Discharged From Rehabilitation by Day Four
Description: % of patients meeting predetermined discharge criteria at 96 Hours post-surgery.
  The discharge criteria were: self dependent (dress, personal care); in and out of bedd independently; up and down stairs; walk with crutches/stick; 80 degrees knee flexion; able to straight leg raise operated limb.
Time Frame: 96 hours
Population: Patients included following randomisation
Measure: Number; unit: percentage of patients
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
percentage of patients | 77 | 82
Statistical Analysis 1: Comparison: Patient Controlled Epidural (PCEA) vs Local Infiltration Analgesia (LIA); Test type: Superiority or Other; p = 0.332, Chi-squared — Significance was set at <0.01

2. Secondary Outcome: Average Post-operative Length of Stay
Description: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Time Frame: Average number of days spent in hospital follwoing surgery, an expected average of 5 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
days | 4 [2 to 20] | 4 [2 to 12]

3. Secondary Outcome: Verbal Rating Score (VRS) Pain Scores
Description: Summary 24 hour Verbal rated numerical pain scores were gathered each day. Scale range 0-10 where 0 is no pain and 10 is worst imaginable pain
Time Frame: 24hours, 48 hours and 72 hours post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
units on a scale
  Theatre Day( asked at 24 hrs) | 3 (4) | 3 (4)
  Post-operative day one( asked at 48hrs) | 3 (3) | 4 (3)
  Post-operative day two(asked 72 hrs) | 3 (2) | 4 (3)

4. Secondary Outcome: Post-operative Urinary Catheterisation Rates
Description: % of patients requiring catheterisation for urinary retention post-surgery
Time Frame: 72 hours post-surgery
Measure: Number; unit: percentage of patients catheterised
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
percentage of patients catheterised | 9.2 | 4.4

5. Secondary Outcome: Post-operative Nausea and Vomiting Scores
Description: percentage of patients reporting either symptoms of nausea or vomiting over the first 72 hours following surgery. Scale 0-2 wherein 0=no nausea and vomiting, 1=nausea and 2= nausea and vomiting
Time Frame: 24hours, 48 hours and 72 hours post-surgery
Measure: Number; unit: percentage of patients reporting PONV
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
percentage of patients reporting PONV | 16 | 14

6. Secondary Outcome: Day of Ambulation
Description: Proportion of patients per day to ambulate for the first time with the physiotherapist > 3 Metres
Time Frame: theatre day, day 1 post-surgery, day two post-surgery
Measure: Number; unit: percentage of patients
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
percentage of patients
  Theatre Day | 35 | 51
  Post-operative day one | 65 | 49
  Post-operative day two | 4 | 0

7. Secondary Outcome: Maximal Flexion Angle of the Operative Knee at Discharge From Rehabilitation
Time Frame: On day of discharge from rehabilitation in-patient care (average 96 hours post surgery)
Measure: Median (Inter-Quartile Range); unit: angle of flexion (degree)
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
angle of flexion (degree) | 80 [60 to 100] | 80 [65 to 105]

8. Secondary Outcome: Patient Reported Outcome Measure - Oxford Knee Score
Description: Units measured on old Oxford Score (12-60) from a 12 point questionnaire. Where in 60 is poor and lower scores are better patient reported outcome scores
Time Frame: one week prior to surgery, 6 weeks post-surgery , one year post-surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
units on a scale
  Pre-operative Oxford Score | 43 [23 to 55] | 43 [20 to 57]
  Six week follow up score | 28 [13 to 53] | 26 [13 to 48]
  One year Follow up score | 19 [12 to 46] | 19 [12 to 54]

9. Secondary Outcome: Total Number of Reported Participants With Complications and/or Adverse Events
Description: The composite number of adverse events reported per group at 30 days and then one year post surgery
Time Frame: 30 days and one year post-surgery
Measure: Number; unit: participants
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Number analyzed (Participants) | 109 | 113
participants
  Reported complications at 30 days | 0 | 2
  Reported complications at one year | 2 | 4

ADVERSE EVENTS:
Time Frame: 30 days post-surgery and one year following surgery
Arm/Group | Patient Controlled Epidural (PCEA) | Local Infiltration Analgesia (LIA)
Serious Adverse Events (participants affected / at risk) | 2/109 | 6/113
Other Adverse Events (participants affected / at risk) | 0/109 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patient Controlled Epidural (PCEA) (N=109) | Local Infiltration Analgesia (LIA) (N=113)
wound Infection at 30 days (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
GI Bleed at 30 days (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction at one year (Cardiac disorders) | 1 (1) | 0 (0)
Wound Infection at one year (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Renal Failure at one year (Renal and urinary disorders) | 0 (0) | 1 (1)
Death at one year (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No